CLINICAL TRIAL: NCT07064798
Title: Evaluating the Use of Limb Cryocompression to Reduce Taxane-induced Peripheral Neuropathy
Brief Title: Cryocompression for CIPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Theresa Jabaley, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-144
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Taxane-Induced Peripheral Neuropathy; CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: Peripheral Neuropathy; Chemotherapy-induced Peripheral Neuropathy; Taxane-Induced Peripheral Neuropathy; CIPN
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Arm A: Cryocompression + Standard of Care Taxane-Based Chemotherapy (Experimental): Participants will be randomized and stratified by chemotherapy regimen and will complete:
  * Baseline visit with questionnaires
  * Standard of care chemotherapy visits with cryocompression
  * End of treatment visit
  Interventions: Device: Paxman Limb Cryocompression System
- Arm B: Standard of Care Taxane-based Chemotherapy (No Intervention): Participants will be randomized and stratified by chemotherapy regimen and will complete:
  * Baseline visit with questionnaires
  * Standard of care chemotherapy visits
  * End of treatment visit

INTERVENTIONS:
Device: Paxman Limb Cryocompression System — An investigational device designed to provide controlled cooling and compression to participant limbs during chemotherapy administration. The device is comprised of a control unit, connecting hose, and two limb wraps. The customizable limb wraps delivers continuous-flow cooling-and-compression to participant extremities
  Other Names: PLCS
  Arms: Arm A: Cryocompression + Standard of Care Taxane-Based Chemotherapy

SUMMARY:
This study aims to evaluate the effectiveness, tolerability, and safety of using cooling therapy and pressure (cryocompression) to reduce peripheral neuropathy, a condition affecting the nerves supplying the arms and legs (limbs) resulting in possible numbness, pain, and/or loss of motor function, that may occur as a result of taxane-based chemotherapy.

The name of the device used in this research study is:

-Paxman Limb Cryocompression System (PLCS)

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness, tolerability, and safety of using cooling therapy and pressure (cryocompression) to reduce peripheral neuropathy, a condition affecting the nerves supplying the arms and legs (limbs) resulting in possible numbness, pain, and/or loss of motor function, that may occur as a result of taxane-based chemotherapy. There is evidence that cooling therapy may be effective for preventing peripheral neuropathy caused by taxane-based chemotherapy.

The U.S. Food and Drug Administration (FDA) has not approved the PAXMAN Limb Cryocompression System as a treatment to reduce peripheral neuropathy.

Participants will be randomized into 1 of 2 groups: Arm A: Cryocompression + Standard of Care Taxane-Based Chemotherapy versus Arm B: Standard of Care Taxane-Based Chemotherapy. Participants will be randomized in a 2:1 manner, meaning a participant is 2 times the chance (approximately 67%) of being in Arm A than in Arm B (approximately 33%). Randomization means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, in-clinic visits, and questionnaires.

It is expected that about 50 people will take part in this research study.

Paxman Coolers, Inc. is providing the Paxman Limb Cryocompression Systems for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Gynecologic or breast malignancy
* Starting 1st cycle of treatment with chemotherapy regimens:

  * Weekly paclitaxel x 12 or weekly paclitaxel/carboplatin x 12 (Breast Oncology)
  * Q3 weeks paclitaxel/carboplatin X 6-8 (GYN)
* Receiving treatment on the main campus of DFCI (these patients are currently seen on Yawkey 9 and 10 and at Chestnut Hill)
* Able to complete questionnaires in English or Spanish

Exclusion Criteria:

* Previous exposure to neurotoxic chemotherapy
* Pre-existing neuropathy
* History of Raynaud's phenomenon, cold agglutinin disease, cryoglobulinemia, cryofibrinogenemia, post-traumatic cold dystrophy, peripheral arterial ischemia, or sickle cell disease
* Undergoing desensitization
* Lymphedema in the limb where the device would be applied
* Open skin wounds or ulcers of the limbs where the device would be applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported CIPN Symptoms Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy module at End of Treatment | Assessed 1-4 weeks after the final taxane infusion (end of treatment).
  Chemotherapy-induced peripheral neuropathy (CIPN) will be assessed using the validated European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy module (EORTC QLQ-CIPN20). This aim is defined as evaluating the incidence and severity of subjectively reported CIPN symptoms, including numbness, tingling, and pain in hands and feet. Clinically significant CIPN is expected to emerge during taxane-based treatment and will be captured at the follow-up visit post-treatment.
Duration of Cryocompression Tolerated During Neurotoxic Chemotherapy | Up to 12 weeks
  Tolerance of cryocompression will be defined by the total amount of time (in minutes) the participant is able to wear cryocompression devices during chemotherapy infusions. This aim evaluates feasibility and tolerability from the patient perspective, based on self-reported ability to continue cryocompression throughout the infusion. Early removal or shortened wear time due to discomfort will be recorded.
Incidence of Core Temperature Decrease >1°F and Skin Intolerance Symptoms Associated with Cryocompression | Throughout each chemotherapy infusion visit when cryocompression is applied. Up to 12 weeks
  This aim assesses the physiological safety of cryocompression. Core body temperature will be monitored orally before, during, and after cryocompression application, with any decreases greater than 1°F considered significant. Skin will be evaluated for intolerance signs (e.g., white or greyish-yellow discoloration, pain, tingling, numbness, or pressure) on cryocompressed limbs. The aim is defined as the absence of these adverse effects during cryocompression use.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Jabaley Leonarczyk, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute; Leonarczyk, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu